CLINICAL TRIAL: NCT02111967
Title: Adequacy of Serum Vitamin B12 Measurement in Type 2 Diabetic Patients Treated With Metformin in Comparison to Holotranscobalamin Measurement
Brief Title: Study to Identify Adequate Biomarker to Detect Vitamin B12 Deficiency in Type 2 Diabetic Patients Treated With Metformin
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Solothurner Spitäler AG (Unknown)
Responsible Party: Principal Investigator, Philipp Walter, PhD, Dr., University of Basel
Other Study IDs: PCRG_Metformin_CMG
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — All blood samples investigated in this study will be destroyed one week after withdrawal. All patient information obtained as a result of the study will be regarded as confidential and made anonymous using a unique study ID number instead of name and surname of the patient.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes mellitus type 2, Metformin: The case group consists of patients with diagnosed diabetes mellitus type 2 treated with Metformin.
  Interventions: Other: Questionnaire administration; Other: Laboratory biomarker analysis
- Diabetes mellitus type 2: The control group consists of patients with diagnosed diabetes mellitus type 2 which do not have metformin treatment
  Interventions: Other: Questionnaire administration; Other: Laboratory biomarker analysis

INTERVENTIONS:
Other: Questionnaire administration
Other: Laboratory biomarker analysis

SUMMARY:
In this study we compare the vitamin B12 status by measuring serum vitamin B12 and holotranscobalamin in type 2 diabetic patients with and without metformin treatment. Afterwars we investigate which biomarker could be adequate to reflect B12 status in metformin-treated patients.

With the help of a questionnaire we assess clinical, nutritional and demographic factors which are associated with vitamin B12 deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM > 6 months
* Metformin treatment for at least 6 months
* Age > 18 years
* Ability to give written informed consent
* No metformin treatment in the last 6 months (control group)

Exclusion Criteria:

* Concurrent intake of preparations containing VB12 (within the last 3 months prior to study participation)
* Lack of written and/or oral understanding in German, French, Italian or English languages
* Diagnosis of Transcobolamin transporter defect
* Diagnosis of Chronic or acute liver diseaseliver insufficiency with CHILD-PUGH scores B and C and acute hepatitis
* Diagnosis of Renal disease (Creatinine-Clearance <60 ml/min)renal insufficiency stadium III, IV and V (KDOQI) and acute renal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus type 2 treated with and without Metformin.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Measurements of serum vitamin B12 and serum holotranscobalamin concentrations | day 3
  VB12, HoloTc

SECONDARY OUTCOMES:
Questionnaire results | day 8
  Clinical, nutritional and demographic factors which are associated with vitamin B12 deficiency should be determined in patients with T2DM.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Prof., Study Chair — Pharmaceutical Care Research Group; Philipp N Walter, Dr., Principal Investigator — Pharmaceutical Care Research Group; Gottfried Rudofsky, Prof. Dr., Study Director — Kantonsspital Olten
Locations (1):
- Pharmaceutical Care Research Group, Basel, Basel, Switzerland